CLINICAL TRIAL: NCT06149390
Title: Observational Clinical Study of Autologous Hematopoietic Stem Cell Transplantation and Chemotherapy as First-Line Consolidation Therapy After Obtaining a Complete Therapeutic Response in T-Cell Lymphoma
Brief Title: ASCT Versus Chemotherapy as First-Line Consolidation Therapy inT-Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Peking University People's Hospital (Other); Ruijin Hospital (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, Liang Huang, Deputy Director, Huazhong University of Science and Technology
Other Study IDs: 2023PHB202-001
Record Dates: First submitted 2023-11-17; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: T-cell Lymphoma Adults
Keywords: NHL; T-cell lymphopma; adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Consoliation with ASCT: consolidation therapy with first-line ASCT in PTCL patients who achieved CR after first-line treatment.
  Interventions: Drug: consolidation with ASCT
- non-ASCT: consolidation therapy without first-line ASCT in PTCL patients who achieved CR after first-line treatment.

INTERVENTIONS:
Drug: consolidation with ASCT — high dose chemotherapy （BCNU, etoposide, cytarabine and melphalan)）and auto stem cells transfusion
  Other Names: consoliation therapy
  Groups: Consoliation with ASCT

SUMMARY:
To compare the effectiveness of autologous hematopoietic stem cell transplantation and chemotherapy as first-line consolidation therapy after obtaining a complete therapeutic response in T-cell lymphoma through a multicenter retrospective real-world study in China.

DETAILED DESCRIPTION:
T-cell lymphoma is characterized by high molecular heterogeneity, high disease aggressiveness, and high chemotherapy resistance rate, and the prognosis is extremely poor. Autologous hematopoietic stem cell transplantation (ASCT) is an important consolidation therapy for patients with T-cell lymphoma who have achieved therapeutic response to chemotherapy, but it is still controversial whether the efficacy of ASCT is significantly better than that of chemotherapy consolidation in patients who have achieved a complete therapeutic response. In this study, the investigators compared the efficacy of ASCT with that of chemotherapy as a first-line consolidation therapy for T-cell lymphoma patients who had achieved a complete therapeutic response in a multicenter real-world study in China. This study included patients with primary T-cell lymphoma diagnosed during 2015-2021 at Shanghai Ruijin Hospital, Peking University People's Hospital, and Wuhan Tongji Hospital, and based on electronic case information, the investigators retrieved the diagnosis, staging, extranodal and bone marrow involvement, and induced and consolidated the efficacy of chemotherapy. The participants were divided into ASCT group and consolidation chemotherapy group according to the consolidation therapy adopted after obtaining complete therapeutic response, and the primary endpoint was adopted as progression-free survival, and the secondary endpoints included overall survival, non-recurrent death, and disease progression/recurrence, so as to explore the efficacy of ASCT and chemotherapy as a first-line consolidation therapy after obtaining a complete therapeutic response in T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of T-cell lymphoma, including, but not limited to, Peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS), Angioimmunoblastic T-cell lymphoma (AITL) , ALK-negative anaplastic large cell lymphoma (ALCL, ALK-negative), Enteropathy-associated T-cell lymphoma (EATL), hepatosplenic T-cell lymphoma (HSTCL), and extranodal NK/T-cell lymphoma (ENKTL )
* 18-75 years old;
* Achievement of a complete response (CR) post-chemotherapy;
* Obtaining a complete response (CR) after chemotherapy;-Consistent follow-up visits post-treatment, with comprehensive follow-up data available;

Exclusion Criteria:

* Initially diagnosed with ALK-positive Anaplastic Large Cell Lymphoma (ALCL, ALK- - -CR was not achieved after treatment;
* Lack of complete follow-up information or lack of consent for follow-up and data collection
* T-cell lymphoma secondary to other malignancies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A preliminary count of approximately 80 patients who received ASCT autologous transplantation and 250 patients who received chemotherapy was conducted as a retrospective cohort study, and all eligible patients were proposed to be included in this study.
Sampling Method: Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
overall survival | through study completion, an average of 2 year
  death as a result of any cause

SECONDARY OUTCOMES:
progression-free survival | through study completion, an average of 2 year
  disease progression or death as a result of any cause
incidence of relapse rate | through study completion, an average of 2 year
  disease relapse
incidence of treatment related mortality rate | through study completion, an average of 2 year
  death without disease progression or relapse

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Mo, Principal Investigator — Peking University